CLINICAL TRIAL: NCT01842711
Title: Exclusive Cumulative Irritation Patch Test (21 Day) With Challenge Patch Application
Brief Title: Cumulative Irritation Patch Test
Status: Completed | Type: Observational
Sponsor: Chattem, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CTTA01-010
Record Dates: First submitted 2013-04-24; First posted 2013-04-30 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Allergy; Irritation; Sensitization
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A Cumulative Patch Test with a Challenge Phase is a test devised to ascertain if a chemical agent or agents have the potential to cause contact irritation or contact allergy in the skin. Allergy is only elicited in immunologically competent individuals who have become sensitized through exposure to the chemical agent at a sufficient concentration and for a sufficient duration of time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must not have any visible skin disease that might be confused with a skin reaction to the test trial;
* Subjects must not be participating in another clinical trial at this facility or any other facility;
* Subjects must be willing to avoid using topical or systemic steroids or antihistamines for at least 7 days prior to trial initiation and during the duration of the trial;
* Subjects must understand and execute and Informed Consent Form;
* Subjects must be capable of understanding and following directions;
* Subjects must be considered reliable;
* Subjects must be aged 16 to 79 years, inclusive;
* Subjects aged less than 18 years must have a parent or legal guardian execute the Informed Consent Form.

Exclusion Criteria:

* Subjects in ill health or taking medications, other than birth control, which could influence the purpose, integrity or outcome of the trial;
* Female subjects who report orally they are pregnant, planning to become pregnant or nursing during the course of the trial;
* Subjects who have a history of adverse reactions to adhesive tape, cosmetics, Over-The-Counter drugs or other personal care products;
* Subjects judged by the PI to be inappropriate for the trial.

Ages: 16 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 240 subjects will be enrolled in the trial so that at least 200 subjects will complete the trial. Subjects who meet all of the inclusion criteria and none of the exclusion criteria will be eligible to enroll into the trial.
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Primary or Cumulative Irritation Potential of the skin | 21 days
  This will be measured by the evaluation of the test sites (skin)by a trained assessor with a predetermined scale for skin irritation.

SECONDARY OUTCOMES:
Allergic Contact Sensitization Potential | 21 days
  After the repeated application period of the test material, a rest period will be employed. The test material will be applied to a naïve site and then will be evaluated by a trained assessor with a predetermined scale for skin irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caswell, PhD, Principal Investigator — Consumer Product Testing Company
Locations (1):
- Consumer Product Testing Company, Inc., Fairfield, New Jersey, United States